CLINICAL TRIAL: NCT02335736
Title: Can Antagonist Protocol be the Protocol of Choice in in Vitro Fertilization Patients?
Brief Title: Antagonist Protocol in IVF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, lecturer of obstetrics and gynecology, Woman's Health University Hospital, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA2015
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: infertility
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal (Active Comparator): Human menopausal gonadotrophin IM daily was administrated from day 2 of the cycle. The Gonadotropins releasing hormone antagonist GnRH ant (Cetrotide, Serono, Geneva, Switzerland) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC.
  Interventions: Drug: Gonadotropins releasing hormone antagonist
- Poor responders (Active Comparator): Human menopausal gonadotrophin IM daily was administrated from day 2 of the cycle. The Gonadotropins releasing hormone antagonist GnRH ant (Cetrotide, Serono, Geneva, Switzerland) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC
  Interventions: Drug: Gonadotropins releasing hormone antagonist
- Polycystic ovarian disease (Active Comparator): Human menopausal gonadotrophin IM daily was administrated from day 2 of the cycle. The Gonadotropins releasing hormone antagonist GnRH ant(Cetrotide, Serono, Geneva, Switzerland) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC
  Interventions: Drug: Gonadotropins releasing hormone antagonist

INTERVENTIONS:
Drug: Gonadotropins releasing hormone antagonist
  Other Names: Cetrotide, Serono, Geneva, Switzerland

SUMMARY:
The antagonist protocol in a novel method of stimulation in the in vitro fertilization (IVF) patients. It has been tried in poor responders, polycystic ovary (PCO) patients and normal females undergoing IVF. Can it be used with the same efficacy in all patients?

ELIGIBILITY:
Inclusion Criteria:

* age: 20- 44 years
* Poor responder females according to Bologna criteria
* Polycystic ovarian disease females according to Rotterdam criteria
* Females with infertility causes other than poor responders, or PCO; male factor or tubal block

Exclusion Criteria:

* refusal to get enrolled in the study
* cases of infertility due to severe male factor

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
number of oocytes collected and fertilized | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt